CLINICAL TRIAL: NCT03073304
Title: A Randomized Controlled Study With the Aim to Compare Crystalloid Prime Solution With a Prime Solution Containing Packed Red Blood Cells in Relation to the Patient's Regional Metabolic Needs and Immunological Influence During Isolated Limb Perfusion
Brief Title: A Randomized Controlled Study Comparing Priming Solution Containing Crystalloid or Packed Red Blood Cells in Patients Treated With Isolated Limb Perfusion.
Acronym: ILP-Prime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILP-Prime
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Melanoma; Sarcoma
Keywords: isolated limb perfusion
MeSH Terms: conditions — Melanoma; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Erythrocyte based prime solution
  Interventions: Drug: Erythrocyte based prime solution
- Intervention (Experimental): Crystalloid based prime solution
  Interventions: Drug: Crystalloid based prime solution

INTERVENTIONS:
Drug: Crystalloid based prime solution — Crystalloid based prime solution
  Arms: Intervention
Drug: Erythrocyte based prime solution — Erythrocyte based prime solution
  Arms: Control

SUMMARY:
The primary aim of this study is to investigate the possibility to replace an erythrocyte based prime solution with a crystalloid based prime solution while maintaining metabolic function. Secondary also to study if potentially reduced immunological influence is obtained during hyper thermic isolated limb perfusion with a crystalloid based prime solution.

ELIGIBILITY:
Inclusion Criteria:

1. The patient scheduled for treatment with isolated hyperthermic perfusion
2. Age over 18 years.
3. Signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-24 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Lactate level during and after perfusion. | 1 hour
  Lactate level during and after perfusion.

SECONDARY OUTCOMES:
Arterial oxygen and regional venous oxygen saturation during and after completion of perfusion. | 1 hour
  Arterial oxygen and regional venous oxygen saturation during and after completion of perfusion.
Hematocrit during and after completion of perfusion. | 1 hour
  Hematocrit during and after completion of perfusion.
Oxygen extraction during, and after perfusion. | 1 hour
  Oxygen extraction during, and after perfusion.
Complications | 30 days
  Serious Adverse Events (SAEs) level III-V within 30 days.
Immunological effects | 30 days
  Changes in proportion of immune cells measured as CD3 + (T cells), CD3 + 4 + (helper T cells), CD3 + 8 + (cytotoxic T cells), CD3 + DR + (activated T cells), CD3 + 4 + 45RA + (naive helper T cells), CD3 + 8 + 45RA + (naïve cytotoxic T cells), CD3 + 4 + 45RO + (helper T cells), CD3 + 8 + 45RO + (cytotoxic memory T cells), CD3-56 + 16 + (NK cells), CD3 + 56 + 16 + (activated T cells), CD5 + (T-cells and some B-cells), CD19 + (B cells), CD5 + 19 + (subset of mature B cells mainly form polyspecific antibodies of the IgM class) will be measured before ILP, after 7 and 30 days post ILP

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corderfeldt Keiller A, Holmen A, Hansson C, Ricksten SE, Bragadottir G, Olofsson Bagge R. Non-invasive and invasive measurement of skeletal muscular oxygenation during isolated limb perfusion. Perfusion. 2023 Jul;38(5):1019-1028. doi: 10.1177/02676591221093201. Epub 2022 May 16. PMID 35575302